CLINICAL TRIAL: NCT02393170
Title: Virtual Reality Intervention for Stroke Rehabilitation - Home Based (Stage 2)
Brief Title: Home-based -Virtual Reality Intervention for Stroke Rehabilitation
Acronym: Home-VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-14-1764-HW-CTIL
Record Dates: First submitted 2015-02-22; First posted 2015-03-19 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- self-training using video-games (Experimental): Participants will receive a video-game console and will be asked to play video-games for one hour a day X 6 days a week for 5 weeks.
  Interventions: Other: self-training using video-games
- traditional self-training (Active Comparator): Participants will receive a manual and kit of a traditional self-training program and will be asked to perform the program one hour a day X 6 days a week for 5 weeks.
  Interventions: Other: traditional self-training

INTERVENTIONS:
Other: self-training using video-games — Individuals will receive a video-game console and will be taught how to play the games.
  They will be requested to play 60 minutes a day for 5 weeks.
  Arms: self-training using video-games
Other: traditional self-training — Individuals will receive a manual and equipment and will be taught how to perform the exercises. They will be requested to perform the exercises 60 minutes a day for 5 weeks.
  Arms: traditional self-training

SUMMARY:
On-going rehabilitation is needed to maintain and improve the weaker upper extremity following stroke. Community rehabilitation programs for stroke individuals in the chronic stage are often difficult to be implement. Consequently, many individuals remain without structured interventional programs. Self-training programs, where individuals can independently continue to exercise at home, might answer this challenge. However, since exercising alone is boring and not motivating, individuals often stop the prescribed exercises and remain inactive. The use of video-games for self-training might answer this challenge.

Therefore, the investigators aimed to assess the feasibility of using video-games for self-training after stroke. Specifically the investigators aim to compare the (1) training time, (2) satisfaction and (3) effectiveness of a self-training program using video-games compared to a traditional self-training program.

DETAILED DESCRIPTION:
This is a single-blind randomized controlled trial with four assessments; two before and two following the 5-week self training intervention.

Individuals are requested to perform the self training (video-games or traditional exercises) 60 minutes a day for 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 36 months after stroke onset
* lived in the community with family or a caregiver
* mild to moderate weakness the affected upper extremity
* without significant cognitive deficit
* able to walk at least 10-meters (with or without assistance).

Exclusion Criteria:

* Other neurological conditions
* Epilepsy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
self-training time | week 9
  Self-training time for the 5-week program as documented on a daily log sheet by the participants in both self-training programs. The mean weekly training hours per week will also be calculated.
Change in Action Research Arm Test | week 0, week 4, week 9, week 13
  change in functional ability of the weaker upper extremity

SECONDARY OUTCOMES:
Change in Box and Block Test | week 0, week 4, week 9, week 13
  Change in dexterity of the weaker upper extremity as assessed by the Box and Block Test
Change in The Functional Reach Test | week 4, week 9, week 13
  Change in standing balance
Daily enjoyment from the self-training | week 9
  For each daily session participants rated their perceived enjoyment (1-5 points).
Change in the Motor Activity Log (MAL) | week 0, week 4, week 9, week 13
  Change in daily use of the weaker upper extremity by using the MAL. This self-report questionnaire generates two seperate scores ranging from 0 to 5, regarding the amount and quality of the weaker upper extremity
Daily exertion from the self-training | week 9
  For each daily session participants rated their perceived exertion (6-20 on the Borg scale). A mean score will be calculated per week.
Satisfaction from the self-training program | week 9
  Satisfaction from the 5-week program and their perceived benefit from the program for improving their weaker upper extremity and balance on a 5-point Likert scale from "not at all" to "very much".

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Rand, OT, PhD, Study Director — Tel Aviv University
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No